CLINICAL TRIAL: NCT05710809
Title: The SaVe Project-Sarcopenia and Vertigo in Aging Patients With Colorectal Cancer
Acronym: SaVe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital - Rigshospitalet, Department of Occupational Therapy and Physiotherapy (Unknown); Copenhagen University Hospital at Herlev (Other); University Hospital Bispebjerg and Frederiksberg (Other); Odense University Hospital, Department of Geriatric Medicine (Unknown); Amager Hospital (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior researcher, Head of research, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-22064206
Record Dates: First submitted 2023-01-16; First posted 2023-02-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer; Oncologic Complications; Comprehensive Geriatric Assessment; Vestibular Rehabilitation; Geriatric Oncology; Sarcopenia; Vertigo; Cancer; Rehabilitation; Exercise; Geriatric; Elderly; Frail; Older Adults; Chemotherapy; Chemotherapy-induced Peripheral Neuropathy; Resistance Training; Balance Training; Postural Stability; Pragmatic Trial; Personal Medicine; Individualised
MeSH Terms: conditions — Colorectal Neoplasms; Sarcopenia; Vertigo; Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator = Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention groups will receive neoadjuvant, adjuvant or first line palliative chemotherapy (for metastatic disease). In addition, all patients will undergo three months' targeted specialized physical group-based exercise and Comprehensive Geriatric Assessment with corresponding interventions
  Interventions: Other: Targeted specialized physical group-based exercise and Comprehensive Geriatric Assessement
- Usual care group (No Intervention): Patients in the usual care groups will receive standard treatment with neoadjuvant, adjuvant or first line palliative chemotherapy (for metastatic disease). If the patients have other health complaints, these will, as current standard procedure, be treated by oncologist or by referral to general practitioner

INTERVENTIONS:
Other: Targeted specialized physical group-based exercise and Comprehensive Geriatric Assessement — Vestibular rehabilitation, balance- and progressive resistance training for three months' three times/week and Comprehensive Geriatric Assessement including corresponding interventions
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn about the cause of dizziness and decline in walking ability in in older adults ≥65 years during chemotherapy treatment for colorectal cancer. Another goal is to investigate if a comprehensive geriatric assessment and three months' specialized physical group-based exercise three times/week can counteract muscle weakness, vertigo, instability, impaired walking balance, and neuropathy

DETAILED DESCRIPTION:
Frequent adverse effects of chemotherapy in older adults are nausea and fatigue, but our research group have discovered a problem with many also suffering from sarcopenia, vertigo, dizziness, and peripheral neuropathy (CIPN) leading to balance and walking impairments causing increased risk of falls. Moreover, these symptoms are often underreported with inadequate awareness among health professionals leading to deficient focus on the need for targeted rehabilitation. A comprehensive geriatric assessment (CGA) can increase the number of frail, older patients completing chemotherapy and CGA-based interventions can decrease chemotherapy toxicity and improve health-related quality of life (HRQoL). Physical exercise has been shown to reduce muscle weakness, vertigo, dizziness, and impaired balance among older adults requiring limited resources. Therefore, this project aims to investigate the effectiveness of CGA and physical exercise to counteract muscle weakness, vertigo, instability, and impaired walking balance, during chemotherapy and to investigate the interaction between vertigo, postural stability and walking performance, and neuropathy and the prevalence of sarcopenia. The activities of specialized physical exercise planned in this intervention will, as hypothesized, result in a change in muscle strength, walking balance, self-perceived balance disabilities/dizziness, and fear of falling along with changes in peripheral nerve function and autonomic function and severity of CIPN which are the outcomes of this study. Accordingly, expectations are that this intervention will affect the HRQoL among older cancer patients with vertigo and walking impairments and reduce the number of falls and hospital admissions leading to a socioeconomic benefit.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of the oncological departments of receiving neoadjuvant, adjuvant or first line palliative chemotherapy for colorectal cancer
* ≥65 years of age at the time of signing the informed consent form
* Able to speak and read Danish, and to provide a signed informed consent form
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2

Exclusion Criteria:

* Chemotherapy treatment within two years and sequelae of neuropathy, or symptoms of dizziness or vertigo, or balance disturbance
* Severe physical disability that hinders physical exercise
* Dementia, psychotic disorders, or other cognitive diseases or conditions that hinder participation in a clinical exercise-based trial
* Inability to sign informed content
* Patients who have had a consultation in the geriatric outpatient clinic within the past six months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index (DGI) | Three months
  Between-group difference in change in walking balance assessed with Dynamic Gait Index (DGI) scored on a 0-24 point total scale. Higher score means better outcome
30 second Sit-to-Stand Test (30STS) | Three months
  Between-group difference in lower limb muscle strength and endurance

SECONDARY OUTCOMES:
Falls | Baseline, two, four, six, eight, ten, twelve, fourteen, sixteen, eighteen, twenty, twenty-two, and twenty-four weeks
  Self-reported falls
Hospital contacts due to falls | Baseline, three and six months
  Hospital contacts due to falls
Balance disabilities/dizziness | Baseline, three and six months
  Changes in self-perceived balance disabilities/dizziness using the patient reported outcome measure Dizziness Handicap Inventory (DHI) scored on a 0-100 point total scale. Higher score means worse outcome
Fear of falling | Baseline, three and six months
  Changes in fear of falling using the patient reported outcome measure Short Falls Efficacy Scale International (Short FES-I) scored on a 0-28 point total scale. Higher score means worse outcome
Health related quality of life | Baseline, three and six months
  Changes in health related quality of life using the patient reported outcome measure EORTC QLQ-C30. The total score is converted to a 0-100 scale. Higher score means better outcome
Peripheral nerve function | Baseline, three and six months
  Changes in peripheral nerve function using biothesiometer mesured in 0-50 volts. Higher volts means worse outcome
Autonomic function | Baseline, three and six months
  Changes in autonomic function using Vagus device
Chemotherapy induced peripheral neuropathy | Baseline, three and six months
  Severity of chemotherapy induced peripheral neuropathy using the patient reported outcome measure EORTC QLQ-CIPN-20. The total score is converted to a 0-100 scale. Higher score means worse outcome
Muscle strength | Baseline, three and six months
  Changes in muscle strength using HUR Leg Press Rehab performance recorder measuring weight in kilograms
Body composition | Baseline, three and six months
  Changes in body composition using DXA
Muscle strength | Baseline, three and six months
  Changes in muscle strength using handgrip test measuring weight in kilograms

OTHER OUTCOMES:
Walking speed | Baseline, three and six months
  Changes in walking speed using 10 meter walk test measuring gaitspeed in meters per second
Postural control | Baseline, three and six months
  Changes in postural control (standing balance) using HUR SmartBalance platform
Vestibular function | Baseline, three and six months
  Changes in peripheral vestibular function using Video Head Impulse Test (vHIT)
Orthostatic blood pressure | Baseline, three and six months
  Changes in orthostatic blood pressure measured from lying to standing and every minute for five minutes
Body composition | Baseline, three and six months
  Changes in body composition using bioimpedance (BIA)
Muscle quality | Baseline and three months
  Changes in muscle quality using ultrasound
Frailty | Baseline
  Presence of frailty using Geriatric-8 (G8) scored on a 0-17 point scale. Higher score means better outcome
Frailty | Baseline
  Presence of frailty using Clinical Frailty Scale (CFS) scored on a 1-9 point scale. Higher score means worse outcome
Activity level | Baseline and three months
  Description of activity level using activity tracker
Cessation of chemotherapy | After 6, 12, and 24 weeks (from baseline)
  Description of cessation of chemotherapy
Prescribed rehabilitation plan | Follow-up at 1, 2, 3, and 5 years
  Recording of exercise through a prescribed rehabilitation plan
Overall survival | Follow-up at 1, 2, 3, and 5 years
  Recording of overall survival
Hospitalisations | Follow-up at 1, 2, 3, and 5 years
  Recording of hospitalisations
Progression of cancer | Follow-up at 1, 2, 3, and 5 years
  Recording of progression of cancer
Recurrence of cancer | Follow-up at 1, 2, 3, and 5 years
  Recording of recurrence of cancer
Biomarkers of sarcopenia and inflammation | Baseline, three and six months
  Biomarkers of sarcopenia and inflammation collected through blood samples. To determine concentration of inflammatory cytokines; High-sensitivity C-reactive Protein (hsCRP), tumour necrosis factor alpha (TNF- α), interleukin 6 (IL6), interleukin 13 (IL-13), and of muscle atrophy and muscle wasting (growth differentiation factor 11 (GDF11), and growth differentiation factor 15 (GDF-15). Blood samples are analysed by standard ELISA-analyses for plasma samples.
Vision | Baseline
  Measurement of vision using a Snellen chart

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Copenhagen University Hospital - Herlev and Gentofte Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Piper KS, Suetta C, Schou JV, Ryg J, Andersen HE, Langevad LV, Evering D, Mikkelsen MK, Lund C, Christensen J. The SaVe project - Sarcopenia and Vertigo in aging patients with colorectal cancer: A study protocol for three randomized controlled trials. J Geriatr Oncol. 2024 May;15(4):101770. doi: 10.1016/j.jgo.2024.101770. Epub 2024 Apr 16. PMID 38631243